CLINICAL TRIAL: NCT06867666
Title: Behavioral Treatment of Insomnia in Active-Duty Service Members With Traumatic Brain Injury
Acronym: CBTBI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Noctem, LLC (Industry)
Collaborators: Naval Health Research Center (U.S. Federal Agency); United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Principal Investigator, Anne Germain, CEO, Noctem, LLC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TP230315
Record Dates: First submitted 2025-02-26; First posted 2025-03-10 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Insomnia; TBI (Traumatic Brain Injury)
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- In-Person CBT-I (Experimental)
  Interventions: Behavioral: In Person CBT-I
- CBT-I via COAST (Experimental)
  Interventions: Behavioral: CBT-I via COAST
- Treatment as Usual (No Intervention): Participants will receive only TBI-related interventions. No insomnia-specific interventions will be provided.

INTERVENTIONS:
Behavioral: In Person CBT-I — 6-week CBT-I delivered in-person at the TBI Clinic at NMCSD or via telehealth on a secure, Health Insurance Portability and Accountability Act (HIPAA) compliant platform by a doctoral-level clinician.
  Arms: In-Person CBT-I
Behavioral: CBT-I via COAST — 6-week CBT-I delivered remotely via a clinician supervised digital platform by a doctoral-level clinician.
  Arms: CBT-I via COAST

SUMMARY:
The objective of the study is to conduct a randomized controlled trial of Cognitive Behavioral Therapy for Insomnia (CBT-I) in a sample of active-duty sailors with a history of traumatic brain injury (TBI). The investigators will test the impact of CBT-I on insomnia symptoms as well as post-concussive symptoms, psychological symptoms, and neurocognitive functioning in comparison to treatment as usual. The investigators will also compare the effectiveness of traditional in-person CBT-I and CBT-I delivered via a clinician-supervised digital health platform, Clinician Operated Assistive Sleep Technology (COAST) in comparison to treatment as usual on symptoms of insomnia, post-concussive symptoms, neurocognitive functioning, and psychological health. Participants will be assessed at baseline, post-treatment, and 3 months later.

ELIGIBILITY:
Inclusion Criteria:

1. Active duty Sailors, activated Reservist Sailors: The study focuses on the treatment in Sailors. Therefore, eligible participants must be active duty Navy, or activated Reservist Navy. Military personnel from other branches, Veterans, other DoD beneficiaries, and civilians are not eligible for the study.
2. Diagnosis of chronic insomnia; PSQI score > 9: The study focuses on the treatment of insomnia. Therefore, eligible participants must have received a diagnosis of chronic insomnia by the study evaluators.
3. History of TBI: The study focuses on the treatment of insomnia in Sailors with TBI. Therefore, eligible participants must have a confirmed history of TBI by the study evaluators.
4. Stable for at least 8 weeks on psychotropic and hypnotic medications: ADSMs currently using prescribed psychotropic and hypnotic medications will be eligible to participate in the trial if they have been on the same medication(s) and at the same dose(s) for at least 8 weeks and there are no expected changes over the course of the acute intervention phase (i.e., up to 6 weeks). Medication usage and changes will nevertheless be tracked prospectively and be considered in the analytical plan should changes occur. To ensure that the three groups are equivalent in composition, the randomization process will be stratified by the use/non-use of psychotropic and hypnotic medication.
5. Stable on continuous positive airway pressure therapy for sleep apnea for at least 90 days and usage of 4 hours or more per night, for at least 70% of the nights: ADSM with comorbid with sleep disordered breathing (SDB) will be eligible to participate in the trial if they are currently stable on continuous positive airway pressure therapy for at least 4 weeks. It is increasingly recognized that insomnia and SDB are often comorbid in military samples56-60. Therefore, exclusion of participants with comorbid SDB would significantly compromise the external validity of the proposed clinical trial. However, SDB requires independent treatment and, if untreated or under-treated comorbid sleep disorder, may be exacerbated by sleep restriction or stimuli control.
6. Own a smart device: Participants in all three treatment delivery conditions will use the COAST app to complete the electronic daily sleep logs and study assessments. Thus, ownership of a smartphone will be required.

Exclusion Criteria:

1. Unable to give informed consent: Individuals who are unable to give informed consent cannot be enrolled in the study. A decisional capacity to consent test, which will be submitted for approval to the Institutional Review Board (IRB), will be used to determine whether a potential participant has the capacity to provide consent on their own behalf.
2. Severe TBI: Individuals with severe TBI will be excluded from this study due to complex medical needs which may require close medical attention and pose safety concerns with regards to completing the study procedures.
3. Potential alcohol use disorder: Individuals who meet diagnostic criteria for current alcohol or substance use disorders will be excluded as these conditions may perpetuate insomnia and daytime impairments and pose safety concerns with regards to completing the study procedures.
4. Inability to comprehend or read English: Participants with demonstrated inability to comprehend or read English will not be eligible for the study. The intervention is highly dependent on understanding the treatment rationale and adhering to behavioral sleep modification instructions. The treatment materials for in-person CBT-I and for CBT-I delivered via digital health platform are only available in English at this time and is the treating clinician's only spoken language. An inability to comprehend or read English limits engagement in CBT-I, and adversely impacts the risk/benefit ratio of participating in the study. Because the study is limited to ADSMs of the United States, it is expected that nearly all potential patients are proficient in reading, writing, speaking, and understanding English, even is English is not their primary language.
5. Serious mental health diagnosis such as bipolar disorder or psychosis; or seizure disorder: Participants who have been previously diagnosed with psychotic or bipolar disorders, or who endorse symptoms of these conditions during the psychiatric assessments, will not be included in the trial because the mild and transient sleep deprivation induced by sleep restriction and stimulus control may exacerbate symptoms and increase the risk of participating in the study. Similarly, individuals with untreated or treatment-resistant seizure disorder will be excluded because seizures may be precipitated or exacerbated by sleep restriction.
6. Hypersomnia disorder: Potential participants that have been diagnosed with hypersomnia that can be exacerbated by the transient and mild sleep deprivation induced by sleep restriction and stimulus control will not be included in the trial as the interventions pose greater safety risks for these participants.
7. Working rotating shifts or requiring that the ADSM report to work earlier than 6am: Potential participants working rotating shifts or who are required to work earlier than 6am will not be included in the trial. Waking up at the same time every day, including on weekends, is a critical aspect of both sleep restriction and stimulus control procedures. Working rotating shifts prohibits participants from adhering to this critical treatment guideline. Being required to work earlier than 6am similarly presents a challenge to waking up at the same time every day, especially on non-workdays when waking earlier than 6am is an unnatural wake time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | The Insomnia Severity Index (ISI) will be administered at the baseline appointment, treatment weeks 2, 4, and 6, within 10 days post-intervention, and the 3-month follow-up to measure insomnia symptoms severity
  The Insomnia Severity Index is a 7-item self-report questionnaire that assesses subjective severity of insomnia symptoms, degree of satisfaction with sleep, nature and noticeability of daytime impairments, and concerns caused by sleep difficulties. Each item is rated on a 0 to 4-point scale. A cut-off score of 14 has been shown to optimize sensitivity and specificity. Scores from 0 to 7 reflect clinically insignificant insomnia; scores from 8 to 14 reflects subthreshold insomnia; scores from 15 to 21 reflect clinically significant insomnia of moderate severity; and scores from 22 to 28 reflect clinically significant, severe insomnia. Reductions of 6 or 8 points or more on the ISI reflect treatment response.
Rivermead Post-Concussion Questionnaire (RPCQ) | The Rivermead Post-Concussion Questionnaire will be administered at the baseline appointment, within 10 days post-intervention, and 3 month follow up appointment
  The Rivermead Post-Concussion Questionnaire will be used to examine post-concussive symptoms. It is a 16-item self-report questionnaire that assesses post-concussive symptoms in the physical, cognitive, and somatic domains. Each symptom is rated on a 5-point scale of 0 = not experienced at all to 4 = a severe problem. The questionnaire has demonstrated good reliability and consistency. It takes approximately 3 minutes to administer. It is recommended by the Department of Defense (DOD) and Department of Veterans affairs (VA) for traumatic brain injury (TBI) research and clinical evaluations. It was previously used as a measure of post-concussion symptoms in a prior trial of CBT-I in a TBI sample demonstrating moderate effects.
Post-Traumatic Stress Disorder Checklist (PCL-5) | The Post-Traumatic Stress Disorder Checklist will be administered at the baseline appointment, within 10 days post-intervention, and 3-month follow up appointment.
  Post-Traumatic Stress Disorder Checklist (PCL-5) is a self-report questionnaire that includes 20 items that correspond to the four symptom clusters of PTSD. Each item is rated on a 5-point scale, ranging from 0 (Not at all) to 4 (Extremely). The sum of item scores rage from 0 to 80, with higher scores indicating more severe PTSD symptoms. It is used extensively in clinical practice and research investigating PTSD in military populations with good psychometric properties. It takes approximately 3 minutes to administer.
Patient Health Questionnaire-8 items (PHQ-8) | The Patient Health Questionnarie-8 items will be done at the baseline appointment, within 10 days post-intervention, and 3-month follow up appointment.
  Patient Health Questionnaire-8 items (PHQ-8) is the depression module of the self-administered version of the Primary Care Evaluation of Mental Disorders diagnostic instrument, the Patient Health Questionnaire (PHQ). The 8 items are based on the DSM-IV diagnostic criteria for depression. Each item is scored from 0 (not at all) to 3 (nearly every day), with higher score indicating greater depressive symptoms. It has demonstrated reliability and validity and takes approximately 3 minutes to administer. In addition, it has been widely adopted by the DOD and VA for research and clinical evaluation and is therefore highly suitable for the current study.
Generalized Anxiety Disorder Screen - 7-items (GAD-7) | The Generalized Anxiety Disorder Screen 7-items will be completed at the baseline appointment, within 10 days post-intervention, and 3-month follow up appointment.
  Generalized Anxiety Disorder Screen - 7-items (GAD-7) is a self-report measure designed to assess severity of symptoms consistent with generalized anxiety disorder based on DSM-IV diagnostic criteria. Response options are "not at all," "several days," "more than half the days," and "nearly every day," scored as 0, 1, 2, and 3, respectively. Higher score indicate worse anxiety symptoms. The Generalized Anxiety Disorder Screen - 7 items has demonstrated adequate validity and reliability. It is a required instrument when sharing data with the NIMH Data Archive and has been widely adopted by the DOD and VA for research and clinical evaluation.

SECONDARY OUTCOMES:
Sleep Diary | Participants will be instructed to complete the daily sleep logs for 1 week after the baseline appointment, every day during the 6-week acute intervention phase, and for 1-week before the 3-month follow up appointment
  The sleep diary consists of a morning and evening log to assess sleep-wake patterns and daytime behavior that may comprise or facilitate sleep (e.g., naps, caffeine use, alcohol consumption, exercise, activation). The morning log is completed upon awakening in the morning and asks questions regarding the time at which the participant went to bed, attempted to fall asleep, duration of nocturnal awakenings, final time out of bed, and total estimated time spent asleep while in bed, and occurrence of disturbing dreams. Visual analog scales also prompt participants to estimate overall sleep quality and restorative quality. The evening portion of the log is completed before bedtime and asks questions about the preceding day including time of naps, exercise, and the consumption of caffeine, alcohol, and tobacco, (and practice of recommended behavioral modifications when applicable).
Brief Fatigue Inventory (BFI) | The Brief Fatigue Inventory will be administered at the baseline appointment, each week during the 6-week acute intervention, within 10 days post-intervention, and 3 month follow up appointment
  Brief Fatigue Inventory (BFI) is a self-report measure assessing fatigue levels and interference with functioning over the previous 24 hours. The nine items are rated from 0 (no fatigue) to 10 (as bad as you can imagine) and higher scores indicate worse fatigue. The measure has good psychometric properties and has demonstrated sensitivity to change in a pilot study of CBT-I in TBI patients.
The World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) | The World Health Organization Disability Assessment Schedule 2.0 will be completed at the baseline appointment, within 10 days post-intervention, and 3-month follow up appointment
  The World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) is a 12-question, self-report questionnaire assessing general health and disability. The WHODAS 2.0 covers six domains: cognition, mobility, self-care, getting along with others, life activities, and participation. Items are rated from "None," "Mild," "Moderate," "Severe," to "Extreme or cannot do," indicating difficulty over the past month. Higher scores indicate greater disability. The WHODAS 2.0 has excellent psychometric properties.

CONTACTS AND LOCATIONS:
Locations (1):
- Naval Medical Center San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Germain A, Wolfson M, Espejo E, Byrd A, Jurick S, Hungerford L, Sitzer T, Healy K, Chinoy E, Sessoms P, Wallace ML, MacGregor A. Behavioral treatment of insomnia in active-duty service members with traumatic brain injury: study protocol for a randomized clinical trial. Trials. 2026 Feb 2. doi: 10.1186/s13063-026-09483-z. Online ahead of print. PMID 41630034